CLINICAL TRIAL: NCT04901806
Title: A Phase 1/2 Study of PBI-200 in Subjects With NTRK-Fusion-Positive Advanced or Metastatic Solid Tumors
Brief Title: Study of PBI-200 in Subjects With NTRK-Fusion-Positive Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor terminated development of PBI-200
Sponsor: Pyramid Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PBI-200-101
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor, Adult; Brain Tumor, Primary; Desmoplastic Small Round Cell Tumor
Keywords: NTRK; NTRK Fusion; Resistance Mutation
MeSH Terms: conditions — Brain Neoplasms; Desmoplastic Small Round Cell Tumor

STUDY DESIGN:
Intervention Model Description: Dose Escalation: Single-subject cohorts will be enrolled initially, until a subject has a Grade 2 or greater adverse event (AE), at which time a 3+3 design will be utilized. Dose escalation will continue until the maximum-tolerated dose (MTD) is reached, or the Recommended Phase 2 Dose (RP2D) is established.
  Cohort Expansion: Two cohorts will be opened to accrual. Cohort A will enroll subjects with a non-brain primary tumor and Cohort B will enroll subjects with a primary brain tumor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental)
  Interventions: Drug: PBI-200
- Phase 2 Cohort Expansion (Experimental)
  Interventions: Drug: PBI-200

INTERVENTIONS:
Drug: PBI-200 — PBI-200 will be administered orally over continuous 28-day cycles

SUMMARY:
This is a first-in-human, open-label, multicenter, dose-escalation, safety, PK, and biomarker study of PBI-200 in subjects with NTRK-fusion-positive advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, open-label, multicenter, dose-escalation, safety, PK, and biomarker study of PBI-200 in subjects with NTRK-fusion-positive advanced or metastatic solid tumors. Phase 1 will also include subjects with NTRK-amplified advanced or metastatic solid tumors or refractory EWSR1-WT1-fusion-positive desmoplastic small round cell tumors (DSRCTs).

Phase 1 is the dose-escalation portion of the study in which the evaluation of safety and tolerability and establishing the RP2D are primary objectives. Once the RP2D has been established, two expansion cohorts will open to accrual, a Non-Brain Primary Tumor cohort and a Primary Brian Tumor cohort.

Although this was intended to be a Phase 1/2 trial, the trial was terminated without proceeding to Phase 2.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has one of the following solid tumors which has progressed on or following at least one systemic therapy regimen administered for advanced or metastatic disease or for which no approved therapy exists:

  * NTRK-fusion-positive, locally advanced (i.e., not amenable to surgical resection) or metastatic solid tumor Note: Subjects with any grade of malignant glioma previously treated with systemic therapy are eligible.

Phase 1

* NTRK-gene amplified, locally advanced or metastatic solid tumor
* EWSR1-WT1-positive DSRCTs.
* Subjects with NTRK-fusion-positive solid tumors other than primary brain tumors must have previously received treatment with a TRK inhibitor, unless the subject does not have access to TRK-inhibitor therapy (e.g., no TRK inhibitor is marketed and available to the subject in the subject's country) or the subject has declined treatment with available marketed TRK inhibitors.
* Subjects with NTRK-gene amplified solid tumors, primary brain tumors or EWSR1-WT1-positive DSRCTs may have received prior treatment with a TRK inhibitor but this is not required.

Phase 2

* Has measurable disease by RECIST v1.1 for subjects with non-brain primary tumors or RANO criteria for subjects with primary brain tumors.
* Subjects with non-brain primary tumors must have previously received treatment with a TRK inhibitor and a documented resistance mutation(s) (e.g., solvent front, gatekeeper or xDFG mutation). Archival tissue from a prior biopsy taken after the subject completed TRK inhibitor treatment but prior to additional systemic therapy may be used to meet this eligibility criterion with Medical Monitor approval.
* Subjects with primary brain tumors may have received prior treatment with a TRK inhibitor but this is not required. Biopsies of brain tumors are not required for eligibility.

Key Exclusion Criteria:

* Cytotoxic chemotherapy, biologic agent, investigational agent, or radiation therapy ≤ 3 weeks prior to the first dose of PBI-200 (6 weeks for nitrosoureas).

  * Subjects with either primary brain tumors or brain metastasis must have completed brain radiation therapy 12 weeks prior to the brain MRI obtained within 4 weeks of the first dose of PBI-200.
* Small-molecule kinase inhibitors or hormonal agents ≤ 14 days and within 5 half-lives prior to the first dose of PBI-200.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Phase 1: Number of patients with AEs | Through study completion, estimated as an average of 36 months
  Severity of AEs will be assessed according to the NCI CTCAE v5.0
Phase 1: Recommended Phase 2 Dose | Approximately 12 months
Phase 2: Cohort A - Overall Response Rate (ORR) | Through study completion, estimated as an average of 36 months
  Assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Phase 2: Cohort B - ORR | Through study completion, estimated as an average of 36 months
  Assessed using Response Assessment in Neuro-Oncology (RANO) criteria

SECONDARY OUTCOMES:
Phase 1: Area under the plasma drug concentration-time curve from 0 to 24 hours after one dose and after 28 doses | 29 days
Phase 1: ORR | Through study completion, estimated as an average of 36 months
  Assessed by RECIST for subjects with non-brain primary tumors and by RANO for subjects with primary brain tumors
Duration of Response (DoR) | Through study completion, estimated as an average of 36 months
  Assessed by RECIST for subjects with non-brain primary tumors and by RANO for subjects with primary brain tumors
Progression-free Survival | Through study completion, estimated as an average of 36 months
  Assessed by RECIST for subjects with non-brain primary tumors and by RANO for subjects with primary brain tumors

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Pyramid Biosciences
Locations (42):
- United States (11):
  - John Wayne Cancer Institute at St. Johns Health Center, Santa Monica, California
  - Stanford Hospital and Clinics, Stanford, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Lake Mary, Florida
  - Sylvester Comprehensive Cancer Center (University of Miami), Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Westchester Medical Center, Hawthorne, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Rigshospitalet, University Hospital of Copenhagen, Copenhagen, Denmark
- France (5):
  - Institut Bergonie, Bordeaux
  - Centre Léon Bérard, Lyon
  - Hopital Europeen Georges Pompidou, Paris
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Dr. Senckenberg Institute of Neurooncology, Frankfurt am Main
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Marienhospital Herne, Herne
- Hong Kong (2):
  - Queen Mary Hospital, Pok Fu Lam
  - Prince of Wales Hospital, Shatin
- Italy (6):
  - Azienda Ospedaliero Universitaria delle Marche, Ancona
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - IRCCS (IEO) Istituto Europeo di Oncologia, Milan
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (5):
  - Seoul National University Bundang Hosptial, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea St. Vincent Hosptial, Suwon, Gyeonggi-do
  - Severance Hosptial, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Soul St. Mary's Hosptial, Seoul
- Spain (5):
  - Hospital Universitari Vall d Hebron, Barcelona
  - ICO l Hospitalet, L'Hospitalet de Llobregat
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital General de Catalunya, Sant Cugat del Vallès
- United Kingdom (2):
  - The Christie, Manchester
  - Royal Marsden Hospital Institute Cancer Research, Sutton

IPD SHARING:
Plan to Share IPD: No